CLINICAL TRIAL: NCT00231725
Title: Complaints Associated With Use of Pre-Filled Pen B When Used by Patients With Type 2 Diabetes on Twice-Daily Insulin Therapy
Brief Title: Complaints Associated With Use of Pre-Filled Pen B With Type 2 Diabetics on Twice-Daily Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 9673; H9D-MC-ITAB
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

INTERVENTIONS:
Drug: insulin lispro injection [rDNA origin] Low Mix

SUMMARY:
Trial of new insulin injection pen called Pre-filled Pen B by type 2 diabetics in take home situations. Patients must use insulin lispro injection [rDNA origin] Low Mix twice daily during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Already on Lilly insulin or beginning insulin therapy
* 25 to 75 years old inclusive

Exclusion Criteria:

* Currently using, or had used during previous month, oral diabetes medication that is NOT approved for use in combination with insulin in patient's country
* More than 3 unexplained episodes of severe hypoglycemia within 6 months prior to trial

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2005-09; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To collect complaint data on the Pre-filled Pen B when used by persons with type 2 diabetes to self-administer insulin in take-home situations for 2 months.

SECONDARY OUTCOMES:
To monitor safety, including all adverse events, hypoglycemia, device-related hypoglycemia, and device-related hyperglycemia
To assess overall patient perception of the device's performance through a patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee, United States
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Requena
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlesbrough, United Kingdom

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com